CLINICAL TRIAL: NCT03154775
Title: Study of Safety and Efficacy of Anti-CD19 Chimeric Antigen Receptor T Cell(C-CAR011) Treatment in Subjects With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma
Brief Title: Study of Safety and Efficacy of C-CAR011 in B-NHL Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBMG-C2017003
Record Dates: First submitted 2017-05-13; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Refractory or Relapsed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR011 (Experimental): Lymphocytes will be transduced with lentiviral vector containing CAR-CD19 gene
  Interventions: Biological: C-CAR011

INTERVENTIONS:
Biological: C-CAR011 — Autologous 2nd generation CD19-directed CAR-T cells, single infusion intravenously at a target dose of 0.5-5.0 x 10^6 anti-CD19 CAR+ T cells/kg
  Other Names: Anti-CD19 Chimeric Antigen Receptor T cell

SUMMARY:
This is a single arm, single-center, non-randomized study to evaluate the safety and efficacy of C-CAR011 therapy in relapsed or refractory B cell Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
This is a single arm, single-center, non-randomized study to evaluate the safety and efficacy of C-CAR011 therapy in relapsed or refractory B cell Non-Hodgkin Lymphoma (NHL). The study will include the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation; Lymphodepleting Chemotherapy), Treatment and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate in this study and signed informed consent
2. Age 18-70 years old, male or female
3. Relapsed or refractory B cell non-Hodgkin's lymphoma

   * 1 Histologically diagnosed as DLBCL(including PMBCL) or follicular lymphoma(grade Ⅲb) according to the NCCN non-Hodgkin's lymphoma Clinical Practice Guidelines (1st edition 2017)

     1. Progressive disease after the last standard chemotherapy regimens
     2. Stable disease after the last standard chemotherapy regimens
     3. Relapsed within 12 months after prior autologous SCT
   * 2 Follicular lymphoma(stage Ⅲ-Ⅳ)(grade Ⅰ-Ⅲa)

     1. At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy
     2. Less than 1 year between last chemotherapy and progression
   * 3 Mantle cell lymphoma

     1. Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT
     2. Disease relapsed or progressed after most recent therapy
     3. Relapsed within 12 months after prior autologous SCT
4. All subjects must have received adequate prior therapy including anti-CD20 monoclonal antibody (unless tumor is CD20-negative) and an anthracycline containing chemotherapy regimen. The standardized treatment regimens reference to NCCN non-Hodgkin lymphoma Clinical Practice Guidelines (2017 Version 1)
5. At least one measurable lesion per revised IWG Response Criteria (the longest diameter of the tumor ≥ 1.5 cm)
6. Expected survival ≥ 12 weeks
7. ECOG score 0-1
8. Adequate pulmonary, hepatic, renal and cardiac function
9. At least 2 weeks from receiving previous treatment (radiotherapy or chemotherapy therapy) prior to leukapheresis,or at least 4 weeks from monoclonal antibody therapy prior to CAR T infusion
10. No contraindications of leukapheresis
11. Female subjects in childbearing age, their serum or urine pregnancy test must be negative, and must agree to take effective contraceptive measures during the trial

Exclusion Criteria:

1. Prior treatment with CAR T therapy or any other genetically modified T cell therapy
2. Relapse after allogeneic hematopoietic stem cell transplantation
3. Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis is allowed), Prophylactic antibiotic, antiviral and antifungal treatment is permissible
4. Hepatitis B or hepatitis C virus infection (including carriers), syphilis, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV-infected people
5. Patients with class III and IV heart failure according to the NYHA Heart Failure Classifications
6. QT interval prolongation≥450 ms
7. A history of epilepsy or other central nervous system disorders
8. No evidence of CNS lymphoma by head enhancement scan or magnetic resonance imaging
9. The patient had a history of other primary cancers, with the following exceptions

   * 1 Excisional non-melanoma such as cutaneous basal cell carcinoma
   * 2 Cured in situ carcinoma such as cervical cancer, bladder cancer or breast cancer
10. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy
11. Used of systemic steroids within two weeks (using inhaled steroids is an exception)
12. Women who are pregnant or lactating or have breeding intent in 6 months
13. Participated in any other clinical trial within three months
14. The investigators believe that any increase in the risk of the subject or interference with the results of the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety(Incidence of adverse events) | 12 weeks
  Incidence of adverse events (AEs)
Objective response rate (ORR) | 12 weeks

SECONDARY OUTCOMES:
Objective response rate (ORR) | 12 months
Duration of remission(DOR) | 12 months
Progression free survival(PFS) | 12 months
Overall survival(OS) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology,Shanghai Tongji Hospital, Tongji University School of Medicin, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided